CLINICAL TRIAL: NCT02514629
Title: Randomized, Double-blind, Parallel, Placebo-controlled, Clinical Trial to Assess the Efficacy of Testosterone, Metformin, or Both, for the Treatment of Obesity-induced Male Hypogonadism
Brief Title: Testosterone, Metformin, or Both, for Hypogonadism in Obese Males
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Fundación Pública Andaluza para la Investigación de Málaga en Biomedicina y Salud (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: CMCS240281
Record Dates: First submitted 2015-07-15; First posted 2015-08-04 (Estimated); Last update posted 2024-12-13 (Actual); Status verified 2024-12

CONDITIONS: Hypogonadism; Obesity
Keywords: Hypogonadism; Obesity; Erectile Dysfunction; Testosterone; Metformin; Weight Loss; Insulin Resistance
MeSH Terms: conditions — Hypogonadism; Obesity; Erectile Dysfunction; Weight Loss; Insulin Resistance | interventions — Metformin; testosterone undecanoate

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- Placebo (Placebo Comparator): Placebo for 52 weeks
  Interventions: Drug: Placebo
- Metformin (Experimental): Metformin 850 mg tablets twice daily for 52 weeks
  Interventions: Drug: Metformin
- Testosterone (Experimental): Testosterone Undecanoate 1000 mg/4ml im injection each 12 weeks for 52 weeks
  Interventions: Drug: Testosterone Undecanoate
- Metformin + Testosterone (Experimental): Metformin 850 mg tablets twice daily + Testosterone Undecanoate 1000 mg/4ml im injection each 12 weeks for 52 weeks
  Interventions: Drug: Metformin + Testosterone Undecanoate

INTERVENTIONS:
Drug: Placebo
  Arms: Placebo
Drug: Metformin
  Other Names: Glucophage; Dianben
  Arms: Metformin
Drug: Testosterone Undecanoate
  Other Names: Nebido; Reandron
  Arms: Testosterone
Drug: Metformin + Testosterone Undecanoate
  Arms: Metformin + Testosterone

SUMMARY:
The purpose of this study is to examine the effects of metformin, testosterone, or both, in males with obesity-related hypogonadism. This study will evaluate changes in insulin resistance, weight loss, body composition, testosterone levels,quality of life and erectile dysfunction.

Obese men will receive diet and physical activity counselling, and be randomised to either testosterone, metformin, a combination of both or placebo

ELIGIBILITY:
Inclusion Criteria:

* Men aged 18 to 50 years.
* BMI > or = 30 kg/m2.
* Total testosterone levels <2.3 ng/ml (<8 nmol/l) or testosterone levels 2.3-3.49 ng/ml (8-12 nmol/l) and free testosterone levels <70 pg/ml.
* LH levels <7.7 mIU / ml.
* No evidence of any other pituitary hormone disruption in morning blood sample (normal concentrations of TSH, FT4, Prolactin, ACTH, cortisol and IGF-1
* Being able to provide informed consent before randomization and agree to comply with all the procedures included in the protocol.

Exclusion Criteria:

* Intolerance/allergy to metformin or testosterone undecanoate.
* Previous diagnosis of diabetes mellitus (HbA1c> 6.5% or fasting glucose> 126 mg/dl or glucose> 200 mg/dl after an oral glucose tolerance test)
* Treatment with oral hypoglycemic agents, insulin or GLP-1 analogs.
* Poor kidney function: serum creatinine> 2.0 mg / dl.
* Previous history of prostate cancer or breast cancer.
* Active cancer of any kind.
* History of liver tumor or acute or chronic liver disease with impaired liver function: total bilirubin> 2.0 mg / dl or GOT levels three times the upper limit of normal.
* Central hypogonadism of organic cause
* Use in the past 12 months of any drug that affects the pituitary-gonadal axis.
* Use of oral testosterone, oral or transdermal within 2 weeks prior to study entry, or any testosterone ester in the last 6 weeks or testosterone undecanoate injection in the 6 months prior to study entry.
* Uncontrolled hypertension (SBP> 160 mmHg or DBP> 100 mmHg) despite adequate antihypertensive therapy.
* HIV infection or known active infection with HBV or HCV.
* Thrombotic or embolic disease.
* Heart disease, kidney or liver disease.
* Epilepsy or migraine not adequately controlled with treatment.
* Hematocrit> 50% in the screening.
* PSA> 4 ng / ml.
* Severe benign prostatic hypertrophy with an IPSS scale score over 19.
* Evidence of drug or alcohol abuse (> 50 g alcohol / day)
* Hematological diseases that produce increased risk of bleeding after intramuscular injection.
* Serious underlying disease that might affect the patient's ability to participate in the study (eg ongoing infection, gastric ulcers, active autoimmune disease).
* Reduced life expectancy (<12 months) by the presence of comorbidities or advanced terminals.
* Participation in another clinical trial within 30 days before study entry.
* Previous diagnosis of hemochromatosis
* Treatment with phosphodiesterase-5 inhibitors: sildenafil, tadalafil or vardenafil

Ages: 18 Years to 50 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 107 (Actual)
Dates: Start 2013-07-04 (Actual); Primary Completion 2016-07-12 (Actual); Study Completion 2016-07-12 (Actual)

PRIMARY OUTCOMES:
Change in Insulin Resistance | Basal-52 weeks
  Insulin resistance will be measured using Homeostasis Model of Assessment for Insulin Resistance index (HOMA-IR index)
  HOMA-IR=FINS*FGLU/22.5

SECONDARY OUTCOMES:
Change in Body Weight | Basal-52 weeks
  Body weight will be measured on a Tanita Multi-Frequency Body Composition Analyzer MC-180MA (Tanita Corporation, Tokyo, Japan) to assess change in body weight over the 52-week intervention period.
Change in Erectile Dysfunction | Basal-52 weeks
  Changes in Erectile Dysfunction will be evaluated with the International Index of Erectile Function (IIEF-5) questionnaire
Change in the Aging Male Symptom (AMS) Scale | Basal-52 weeks
  Change from baseline on the total score of the AMS rating scale
Change in the Androgen Deficiency in the Aging Male (ADAM) Questionnaire | Basal-52 weeks
  Change from baseline on the ADAM Questionnaire
Change in Testosterone Levels (Total and Free) | Basal-52 weeks
  The change from baseline to week 52 in free testosterone and total testosterone levels will be assessed
Change in Body Composition (Fat and Lean Mass) | Basal-52 weeks
  Body Composition will be measured on a Tanita Multi-Frequency Body Composition Analyzer MC-180MA (Tanita Corporation, Tokyo, Japan) to assess changes in body composition (fat mass, lean mass, total body water) over the 52-week intervention period.
Change in Biochemical Markers of Bone Turnover | Basal-52 weeks
  Change in Bone turnover, measured by serum procollagen type I N-terminal propeptide (PINP) and Beta-CrossLaps (β-CTx)
Change in Metabolic Hormones | Basal-52 weeks
  Changes in Leptin, adiponectin, betatrophin and kisspeptin levels

CONTACTS AND LOCATIONS:
Overall Officials: Jose Carlos Fernandez-Garcia, MD, Principal Investigator — Hospital Universitario Virgen de la Victoria. Malaga
Locations (1):
- Hospital Uiversitario Virgen de la Victoria, Málaga, Malaga, Spain